CLINICAL TRIAL: NCT04569188
Title: Real-time Evaluation of Safety and Efficacy of Convalescent Plasma Units Transfused to Elderly Patients With COVID-19
Brief Title: Convalescent Plasma in COVID-19 Elderly Patients
Acronym: RESCUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale di Mantova (Other)
Responsible Party: Principal Investigator, Massimo Franchini, Director Immunohematology and Transfusion Service, Azienda Socio Sanitaria Territoriale di Mantova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Asstmantova
Record Dates: First submitted 2020-09-04; First posted 2020-09-29 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- convalescent plasma (Experimental): Cohort of elderly patients treated with convalescent plasma
  Interventions: Biological: Convalescent plasma

INTERVENTIONS:
Biological: Convalescent plasma — COVID-19 elderly patients treated with convalescent plasma

SUMMARY:
The trend of the spread of the COVID-19 pandemic demonstrates in Lombardy, starting from 28.03.2020, a slowdown in the exponential phase of infections and the probable reaching of a plateau phase.

However, a marked increase in infections was observed in the so-called "protected structures" such as nursing homes (RSA), both in health staff and in the residents of such facilities. The observed percentage of lethality, according to the more recent data provided by the National Institute of Health, is very high especially among residents.

For these reasons, the city Hospital (ASST) of Mantua , already involved in the use of hyperimmune plasma as a therapy for COVID-19, designed this study in order to evaluate RSA patients and to identify the cases eligible for this treatment.

DETAILED DESCRIPTION:
For a detailed description of the study, see the attached protocol

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (> 65 years old) with SARS-CoV-2 RT-PCR positivity on nasal swab or score higher than 5 with the following characteristics:

  * New onset or worsening of recently onset respiratory symptoms (<10 days);
  * Radiological imaging (CT, X-ray, Ultrasound) of bilateral pulmonary opacities not fully explained by pleural effusion, pulmonary or lobar atelectasis, pulmonary nodules;
  * Respiratory failure (SpO2 <95%) not fully explained by heart failure or water overload (after excluding hydrostatic causes of edema in the absence of risk factors by objective assessment, for example ultrasound);
* Patients who have signed informed consent.

Exclusion Criteria:

* New onset or worsening of respiratory symptoms that began more than 10 days ago;
* Patients with proven hypersensitivity or allergic reaction to plasma, blood products or immunoglobulins;
* Manifest desire not to be included in the research protocol.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Death | 15 days
  Death from any cause

SECONDARY OUTCOMES:
Viral load | 7 days
  Naso-pharyngeal swab

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Franchini, Principal Investigator — ASST Mantova
Locations (1):
- Transfusion Service, Mantova, Italy

REFERENCES:
- [Derived] Franchini M, Glingani C, Morandi M, Corghi G, Cerzosimo S, Beduzzi G, Storti A, Di Stasi V, Rastrelli G, Vignozzi L, Mengoli C, Garuti M, Beccaria M, Inglese F, Caruso B, Petilino RA, Amato M, Nicchio M, Pagani M, Bellani A, Castelli G, Casari S, De Donno G. Safety and Efficacy of Convalescent Plasma in Elderly COVID-19 Patients: The RESCUE Trial. Mayo Clin Proc Innov Qual Outcomes. 2021 Apr;5(2):403-412. doi: 10.1016/j.mayocpiqo.2021.01.010. Epub 2021 Feb 8. PMID 33585799

DOCUMENTS (1):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT04569188/Prot_001.pdf